CLINICAL TRIAL: NCT05020379
Title: Investigation of The Effects of The Erector Spinae Plane Block on The Quality Of Recovery After Laparoscopic Bariatric Surgery: A Prospective Randomized Trial
Brief Title: The Effects of Erector Spinae Plane Block on Bariatric Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-2021/05
Record Dates: First submitted 2021-08-21; First posted 2021-08-25 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Laparoscopic Bariatric Surgery
Keywords: Barıatrıc Surgery.; Erector spinae block; Quality of recovery (QoR-40)

STUDY DESIGN:
Intervention Model Description: Randomized Intervention Model: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (Sham Comparator): The patients in Group N will not receive any intervention. Patients will receive standard multimodal analgesia comprising paracetamol, tenoxicam, and tramadol. The pain intensity will be evaluated with the 0-10 Numeric Rating Scale (NRS). NRS are the simple and most commonly used scales.11 The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."
  Interventions: Procedure: Perioperative and postoperative multimodal analgesia
- Group ESPB (Experimental): The patients in the group ESPB will be placed in sitting pozition. A convex probe ultrasound transducer will be place in a longitudinal parasagittal orientation about 3 cm lateral to spinous process. Local anesthetic (20 ml 0.25% bupivacaine) will be injected bilaterally into the fascial plane on the deep aspect of erector spinae muscle. Standard perioperative and postoperative analgesia protocol will be given and postoperative pain levels will be determined by Numerical rating scale (NRS)
  Interventions: Procedure: Perioperative and postoperative multimodal analgesia; Procedure: ESP Block

INTERVENTIONS:
Procedure: Perioperative and postoperative multimodal analgesia — Patients will receive standard multimodal analgesia comprising paracetamol, tenoxicam, and tramadol.
  The pain intensity during rest and motion will be evaluated with the 0-10 Numeric Rating Scale (NRS). NRS scores for pain and postoperative opioid consumption will be evaluated at 15th and 30th minutes, 1st, 2nd, 6th, 12th, 24th hours, 2nd day.
  Other Names: Global Quality of Recovery-40 score; Standard Pain Follow up
Procedure: ESP Block — Patients in the ESPB group will be placed in a sitting position. A convex probe ultrasound transducer will be placed in a longitudinal parasagittal orientation approximately 3 cm lateral to the spinous process. Local anesthetic (20 ml 0.25% bupivacaine) will be injected bilaterally into the fascial plane on the deep face of the erector spinae muscle. Standard perioperative and postoperative analgesia protocol will be given and postoperative pain levels will be determined by Numerical Rating Scale (NRS). NRS scores for pain and postoperative opioid consumption will be evaluated at 15th and 30th minutes, 1st, 2nd, 6th, 12th, 24th hours, 2nd day.
  Other Names: Global Quality of Recovery-40 score; Standard Pain Follow up
  Arms: Group ESPB

SUMMARY:
The erector spinae plane block (ESPB) is a new technique that is increasingly used in the treatment of acute and chronic pain. Bariatric surgery is a surgical treatment method used in the treatment of morbid obesity and related comorbidities. Providing pain control in obese patients is a topic that remains up-to-date. Poorly controlled early postoperative pain impairs quality of recovery, increases the risk of postoperative pulmonary complications, and is a risk factor for the subsequent development of chronic pain. Therefore, optimizing acute postoperative analgesia is a priority in patients undergoing bariatric surgery. The primary aim of this prospective, randomized study is to evaluate the effect of ESPB on quality of recovery with the QoR-40 questionnaire in patients undergoing elective Laparoscopic Bariatric Surgery.

DETAILED DESCRIPTION:
In the operating room, all patients will receive standard monitoring, including electrocardiography, non-invasive blood pressure, and peripheral oxygen saturation. Patients in the ESPB group will be placed in a sitting position. A convex probe ultrasound transducer will be placed in a longitudinal parasagittal orientation approximately 3 cm lateral to the spinous process. The needle tip was advanced until it will be located in the inter-fascial plane deep to the erector spinae muscle group and superior to the transverse process. Once in position, bupivacaine 0.25%, 20 ml was injected under ultrasound, guidance. The same procedure will be repeated on the contralateral site. Standard perioperative and postoperative analgesia protocol will be given and postoperative pain levels will be determined by Numerical Rating Scale (NRS). NRS scores for pain and postoperative opioid consumption will be recorded on the 15th,30th minute, 1st, 2nd, 12th, 24th hour, 2nd day. Quality of recovery-40 (QoR-40) scores will be given on the ward, at postoperative 24th hour, 3rd and 7th day ( the 3rd and 7th-day scores will be calculated after telephone interview if the patient will be discharged from the hospital).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective laparoscopic bariatric surgery

Exclusion Criteria:

* a history of allergy to local anesthetics
* known coagulation disorders
* infection near the puncture site
* Chronic opioid intake
* Patient with psychiatric disorders
* Can not communicate in Turkish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery (QoR-40) score | postoperative 24th hour
  QoR-40, a 40-item questionnaire that provides a global score and subscores across five dimensions: patient support, comfort, emotions, physical independence, and pain. Each item is rated on a scale of 1-5, providing a minimum score of 40 and maximum of 200. The increase in scores show high quality of recovery.

SECONDARY OUTCOMES:
Postoperative pain: numeric rating scale (NRS) | Postoperative 48 hour
  NRS use numbers to rate pain from 0 (no pain) to 10 (worst pain). Postoperative pain levels will be determined by Numeric Rating Scale (NRS) system
Analgesic consumption | Postoperative 48 hour
  Total opioid consumption at the postoperative period
Side effects | 24 hours
  Rate of side-effect occurrences (such as rate of vomiting,nausea,dizziness)
Sedation score | Postoperative 48 hour
  Evaluation of the level of sedation in patients with a 4-point scale (0=wake, 1=sleepy, easy to verbally arouse, 2=drowsy, 3=does not open their eyes to verbal commands).
mobilization time | Postoperative 24 hour
  The time after surgery to the mobilization of the patient
Quality of Recovery (QoR-40) score | Postoperative 3rd and 7th days
  QoR-40, a 40-item questionnaire that provides a global score and subscores across five dimensions: patient support, comfort, emotions, physical independence, and pain. Each item is rated on a scale of 1-5, providing a minimum score of 40 and maximum of 200. The increase in scores show high quality of recovery.
Postoperative complications | Postoperative 30 days
  Postoperative complications will be identified by visiting patients every day or alternate day during their in hospital course, suplemented by patients medical records using our hospital's electronic patient record database. We will use the Claviene Dindo Classification system from which CC is derived. We defined a postoperative complication as any deviation from the ideal postoperative course, not inherent in the procedure itself and does not constitute a failure to cure. CCI scores willbe calculated using the online CCI calculator.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Basaran, MD, DESA, Study Director — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

REFERENCES:
- [Derived] Toprak H, Basaran B, Toprak SS, Et T, Kumru N, Korkusuz M, Bilge A, Yarimoglu R. Efficacy of the Erector Spinae Plane Block for Quality of Recovery in Bariatric Surgery: a Randomized Controlled Trial. Obes Surg. 2023 Sep;33(9):2640-2651. doi: 10.1007/s11695-023-06748-3. Epub 2023 Jul 24. PMID 37488349